CLINICAL TRIAL: NCT00794053
Title: The Role of Sentinel Lymph Node Biopsy (SLNB) In the Management of Differentiated Thyroid Cancer
Brief Title: The Usefulness of Staining Lymph Nodes During Operations for Cancer Thyroid in Detecting the Nodes That Have Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Yasser Hamza, UAlexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UAlexandria
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Thyroid Cancer; Lymph Node Metastasis
Keywords: Sentinel lymph node; thyroid cancer; neck dissection
MeSH Terms: conditions — Thyroid Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study group (Experimental): The members in this group will undergo intervention by having surgery and lymph node detection by dye staining
  Interventions: Procedure: detecting lymph node metastasis by staining

INTERVENTIONS:
Procedure: detecting lymph node metastasis by staining — this started by collar incision, development of sub-platysmal skin flaps and separation of strap muscles in the midline. This was followed by exposure of the thyroid gland; identification of the thyroid tumour; injection of the dye into the tumour; waiting for the dye to reach the lymph nodes; identifying the stained node; labeling it as the sentinel node (SLN); performing total thyroidectomy and bilateral central neck dissection.
  Other Names: sentinel lymph node detection; staging of thyroid cancer

SUMMARY:
Detection of lymph nodes starting to be involved by cancer spreading from the thyroid gland during operation is useful. It saves the patient from having a second operation to remove these nodes later on when they become obvious. The problem is that there are many lymph nodes around the gland. The theory is that only one node will get the first spill of the tumour cells.

In this study the investigators are trying to use an inert colored material to inject into the tumour. This should run in the same path as the tumour cells and should therefore stain the one lymph node that will be affected first should the tumour spread.

The stained lymph node is excised and examined instantaneously for tumour affection. If it is found to be affected by the tumour, then the operation is extended to include removal of all its fellow lymph nodes. If it is found to be free from the tumour, then this patient does not have tumour spread.

DETAILED DESCRIPTION:
The study includes 45 consecutive patients diagnosed as differentiated thyroid cancer by clinical examination and/or fine needle aspiration cytology (FNAC).

Exclusion criteria are: previous neck surgery, pregnancy and known hypersensitivity to the dye used.

An informed consent was obtained from all the patients. Peroperative workup includes history taking, clinical examination, relevant laboratory investigations including thyroid hormone assay, ultrasonography of the neck with special emphasis on the thyroid focal lesion and cervical lymph nodes. FNAC was attempted in all patients.

All patients were then subjected to operation:

A systematized surgical approach was adopted for the purpose of the study: this started by collar incision, development of sub-platysmal skin flaps and separation of strap muscles in the midline. This was followed by exposure of the thyroid gland; identification of the thyroid tumour; injection of the dye into the tumour; waiting for the dye to reach the lymph nodes; identifying the stained node; labeling it as the sentinel node (SLN); performing total thyroidectomy and bilateral central neck dissection.

The resected specimen was fixed by formaldehyde, stained with hematoxylin and eosin and examined with light microscopy.

If the SLN was found to be free of malignant deposits, it was further examined by immunohistochemical staining.

Statistical analysis: Descriptive statistics were used to analyze demographic data. Sensitivity, specificity and predictive value of the SLN were calculated.

The histopathological report of the excised specimen was considered the criterion standard.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed to have differentiated thyroid carcinoma and has no detectable cervical lymphadenopathy.

Exclusion Criteria:

* Previous neck surgery, pregnancy and known hypersensitivity to the dye used.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-12; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The lymph nodes around the thyroid tumour will be removed and examined under microscopy in all study subjects to verify that the stained node is a true representative to the state of lymph nodes as regards tumour spread | the lymph nodes removed during the surgery will be examined the next day of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Yasser M Hamza, A Professor, Principal Investigator — University of Alexandria
Locations (1):
- Alexandria University Hospitals, Alexandria, Alexandria Governorate, Egypt